CLINICAL TRIAL: NCT05247788
Title: Impaired Risk Awareness During Intoxication in DUI Offenders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mark Fillmore (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Mark Fillmore, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 60239; R01AA028447 (NIH)
Record Dates: First submitted 2022-02-05; First posted 2022-02-21 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Alcohol Use
Keywords: Social drinker
MeSH Terms: conditions — Alcohol Drinking | interventions — Blood Alcohol Content; Bacitracin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intoxicated risk awareness training session (Experimental): Participants will complete an intoxicated risk awareness training session in which they receive a controlled alcohol dose with structured feedback and training to accurately appraise the impairing effects of alcohol and estimate their blood alcohol concentration (BAC).
  Interventions: Behavioral: Blood alcohol concentration (BAC) discrimination training; Behavioral: Performance feedback training
- Alcohol exposure only (Active Comparator): Participants assigned to the alcohol-exposure-only condition undergo the same alcohol dose exposures over the session but receive a general body scan and do not receive feedback concerning BAC or performance.
  Interventions: Behavioral: Blood alcohol concentration (BAC) discrimination training for controls

INTERVENTIONS:
Behavioral: Blood alcohol concentration (BAC) discrimination training — Subjects will receive 0.65 g/kg alcohol to yield a peak BAC of 85 mg/dl (0.085%). They will be trained to accurately estimate their BAC using the Body Scan Exercise with BAC feedback.
  Arms: Intoxicated risk awareness training session
Behavioral: Performance feedback training — This training element targets the driver's self-efficacy by increasing their awareness of the behavioral impairing effects of alcohol that are experienced at BACs at and even below the legal limit (50-80 mg/dl).
  Arms: Intoxicated risk awareness training session
Behavioral: Blood alcohol concentration (BAC) discrimination training for controls — Subjects will receive 0.65 g/kg alcohol to yield a peak BAC of 85 mg/dl (0.085%). They will be given a general Body Scan Exercise with no feedback.
  Arms: Alcohol exposure only

SUMMARY:
This study aims to test the efficacy of experiential-based training to increase DUI offenders' perceptions or risk associated with alcohol use.

DETAILED DESCRIPTION:
This project examines the efficacy of a laboratory-based intervention to increase risk awareness of DUI offenders during states of acute alcohol intoxication. The proposed research will test the efficacy of an innovative experiential-based training approach to improve DUI offenders' ability to appraise their level of intoxication and enhance their risk awareness. DUI offenders will undergo experiential-based training in which they are administered a controlled dose of alcohol and receive structured feedback and mindfulness-based training to accurately appraise the impairing effects of alcohol and estimate their breath alcohol concentration. The research tests the hypothesis that the experiential training will increase DUI offenders' risk awareness in the intoxicated state as evident by reduced disinhibition and risk-taking behavior in response to alcohol, and reduced self-reported alcohol consumption over a follow up period.

A total of 60 DUI offenders and 60 non-offender controls will be recruited. The study tests the degree to which acute alcohol intoxication impairs key indicators of risk awareness in DUI offenders and the efficacy of experiential feedback to increase risk awareness during intoxication. Two key indicators of impaired risk awareness will be assessed during intoxication: 1) increased disinhibition/risk-taking and; 2) reduced perception of intoxication. Two main hypotheses are tested. Hypothesis 1: Prior to training, DUI offenders will display greater disinhibition/risk-taking and less perceived impairment in response to alcohol compared with controls. Hypothesis 2: Experiential feedback training will increase intoxicated risk awareness among DUI offenders as evident by reduced disinhibiting and risk-taking effects in response to alcohol and increased perception of impairment and accuracy of BAC estimation. Offenders and controls will undergo a pre-training assessment of their responses to a controlled dose of 0.65 g/kg alcohol versus a placebo on the two key indicators of risk awareness: disinhibition/risk-taking and perceived intoxication. Experiential feedback training sessions will begin within one week of completing the pre-training assessment of intoxicated risk awareness. Subjects will attend two training sessions in which they are administered a controlled dose of alcohol and receive structured training to accurately estimate their breath alcohol concentration and accurately appraise the behavioral impairing effects of alcohol. Half of the DUI offenders (20 men and 10 women) will be randomly assigned to the training condition and the other half assigned to an alcohol-exposure-only "control" condition. Non-offender, control subjects will undergo the same group assignment procedure. After completing the two training sessions all subjects will be re-tested on the two indicators of risk awareness in response to 0.65 g/kg alcohol: disinhibition/risk-taking and perceived intoxication. The post-training assessment of alcohol responses is identical to the pre-training assessment and will be conducted at 2 time points: 1-week post-training and 3 months post-training, to evaluate retention effects. Alcohol consumption also will be assessed at monthly intervals over the 3 month follow-up to evaluate the training efficacy to reduce high-risk patterns of consumption (e.g., binge episodes).

ELIGIBILITY:
Inclusion Criteria:

* Valid driver's license for at least 5 years
* Drive regularly (weekly basis)

Exclusion Criteria:

* History of physical or psychiatric disease
* Pregnancy
* Breastfeeding
* Substance use disorder (other than nicotine or caffeine use)

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Change in alcohol consumption | Baseline to follow up [Monthly], up to 3 months
  Alcohol consumption will be assessed at monthly intervals from baseline to follow up and will be measured using a timeline follow back assessment. Participants will self-report data on number of days when the participant demonstrates binge drinking (5+ drinks per day for men; 4+ drinks per day for women).
Change in tonic alcohol cravings | Baseline to follow up [Monthly], up to 3 months
  Change in tonic alcohol cravings will be assessed using the Penn Alcohol Craving Scale (PACS) which is a five-item self-report indicated with strong psychometrics that measures the frequency, intensity, and duration of thoughts about drinking over the past week. PACS uses a 0-6 point Likert scale where a higher number higher cravings. Total scores range from 0 to 30.
Change in subjects perceive improvement in their interoceptive ability | Baseline to follow up [Monthly], up to 3 months
  Change in subjects perceive improvement in their interoceptive ability will be assessed by the Multidimensional Assessment of Interoceptive Awareness Ver. 2 (MAIA-2) is a 37-item self-report measure of eight dimensions of self-perceived interoceptive ability. MAIA-2 uses a 0-5 point Likert scale (0=never, 5=always) where higher values indicate a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Fillmore, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

DOCUMENTS (1):
  • Informed Consent Form (2024-07-11): https://cdn.clinicaltrials.gov/large-docs/88/NCT05247788/ICF_000.pdf